CLINICAL TRIAL: NCT01282411
Title: Anatomic Outcomes Following Ozurdex Injection
Brief Title: Anatomic Outcomes Following Ozurdex Injections
Status: Completed | Type: Observational
Sponsor: Barnes Retina Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Rhonda Weeks, Gaurav K. Shah, MD, Barnes Retina Institute
Other Study IDs: 2010.006
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Retinal Vein Occlusions
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Ozurdex(TM) has recently been FDA approved for use in macular edema secondary to retinal vein occlusion. It remains unclear how quickly the drug works and for how long as the initial studies did not have frequent anatomic monitoring. This study will utilize frequent Spectral domain OCT imaging to better understand the onset of treatment effectiveness and duration of action on the anatomic thickness of the retina, in addition to distinguishing structural abnormalities of responders from non-responders.

DETAILED DESCRIPTION:
Focal laser therapy has been the gold standard for the treatment of macular edema secondary to branch vein occlusion (BRVO), though it has not been shown to be effective for central vein occlusion (CRVO). Intravitreal corticosteroids have been shown in many case series to be effective at diminishing macular edema secondary to both BRVO and CRVO. Sustained drug delivery models have been sought after to relieve the need for frequent injections. Ozurdex has recently been found to be effective for the treatment of macular edema following BRVO or CRVO and has been approved by the FDA for these indications. The onset of effectiveness and duration of action on the anatomic thickness of the retina have not yet been demonstrated. In addition, it is uncertain as to when the clinician can label the patient as a responder or nonresponder. We also believe this study will help identify patients that may need more frequent dosing schedules.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with BRVO/CRVO who are otherwise eligible to receive treatment with Ozurdex (TM)

Exclusion Criteria:

* Patients younger than 21 years of age, unwilling or unable to grant informed consent, participation in a clinical trial within the 30 days prior to enrollment. Patients receiving any other ocular therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Branch retinal vein occlusion (BRVO) Central retinal Vein occlusion (CRVO)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav K Shah, MD, Principal Investigator — Barnes Retina Institute
Locations (1):
- Barnes Retina Institute, St Louis, Missouri, United States